CLINICAL TRIAL: NCT01590433
Title: A Prospective Study of Patterns, Predictors, and Mechanisms of Weight Loss With Exenatide Treatment in Overweight and Obese Women Without Diabetes
Brief Title: Weight Loss With Exenatide Treatment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Jody Dushay (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor-Investigator, Jody Dushay, Assistant Professor of Medicine, Beth Israel Deaconess Medical Center
Organization: Beth Israel Deaconess Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2011P000310
Record Dates: First submitted 2012-02-24; First posted 2012-05-03 (Estimated); Results first posted 2020-02-12 (Actual); Last update posted 2021-06-23 (Actual); Status verified 2021-06

CONDITIONS: Obesity
Keywords: Obesity; Overweight; Exenatide; Diet; Women
MeSH Terms: conditions — Obesity; Overweight | interventions — Exenatide; Nutrition Assessment

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Exenatide (Experimental): Subjects will be randomly assigned to the exenatide study treatment group or to the placebo study treatment group. Subjects will have a 33 percent chance of being assigned to the placebo study treatment group and a 66 percent chance of being assigned to exenatide study treatment. Subjects will not be able to choose the study group to which they will be assigned. All study participants will receive individualized dietary counseling based on food logs. Subjects who receive exenatide will not be assigned to follow a reduced-calorie diet in addition to study treatment. Subjects will not know whether they are receiving exenatide or placebo, but the unblinded members of study team will know which they are receiving.
  Interventions: Drug: Exenatide
- Placebo (Placebo Comparator): Subjects will be randomly assigned to the exenatide study treatment group or to the placebo study treatment group. Subjects will have a 33 percent chance of being assigned to the placebo study treatment group and a 66 percent chance of being assigned to exenatide study treatment. Subjects will not be able to choose the study group to which they will be assigned. All study participants will receive individualized dietary counseling based on food logs. Subjects who receive placebo will be assigned to follow a reduced-calorie diet in addition to study treatment. Subjects will not know whether they are receiving exenatide or placebo, but the unblinded members of the study team will know which they are receiving.
  Interventions: Drug: Placebo; Behavioral: Dietary counseling

INTERVENTIONS:
Drug: Exenatide — Subjects will inject 5mcg of exenatide subcutaneously 15 minutes before the morning and evening meal for the first 2 weeks of the study. At study week 2, subjects will increase to 10mcg twice daily for the remainder of the study.
  Arms: Exenatide
Drug: Placebo — Subjects will inject 5mcg of identically dispensed placebo subcutaneously 15 minutes before the morning and evening meal for the first 2 weeks of the study. At study week 2, subjects will increase to 10mcg twice daily for the remainder of the study.
  Arms: Placebo
Behavioral: Dietary counseling — All subjects will also receive individualized dietary counseling. Subjects in the placebo group will be counseled to follow a hypocaloric diet.
  Arms: Placebo

SUMMARY:
The investigators are conducting a study that will investigate the possible mechanisms of weight loss associated with exenatide treatment and the metabolic characteristics of high responders (i.e. subjects who achieve greater than 5% weight loss) to exenatide treatment. The investigators will also examine the magnitude and duration of weight loss among a cohort of high responders over 52 weeks of treatment, and at 3 and 6 months following treatment.

Hypothesis:

The mechanisms of weight loss with exenatide are not fully understood, and weight loss responses to exenatide are highly variable, possibly reflecting distinct metabolic parameters. By identifying and following a group of obese women who lose greater than 5% body weight after short-term exenatide treatment, the investigators can gain insights into the possible mechanisms of weight loss and assess long-term weight loss with this pharmacotherapeutic intervention.

DETAILED DESCRIPTION:
Primary Outcomes

The primary objectives of this study is:

- To investigate possible mechanisms and patterns of weight loss with exenatide treatment, especially among individuals who have robust early weight loss (greater than 5% weight loss in 12 weeks) with exenatide.

Secondary Outcomes

Our secondary objective is to identify metabolic characteristics that predict robust response to exenatide treatment.

Outcome measurements:

* Weight
* Body composition
* Resting energy expenditure (REE)
* Mixed meal test
* Thermic effect of food
* Serum metabolic parameters
* Hunger/Nausea/Satiety visual analog scales (VAS)
* Physical activity monitoring

Study Population

The study population will be generally healthy, non-diabetic women age 18-70 years with BMI 28-48 kg/m^2.

ELIGIBILITY:
Inclusion Criteria:

* Females age 18-70
* BMI 28-48 kg/m^2
* Stable weight (greater than 3 kg weight gain or loss within 6 months of screening visit).
* Ability to give informed consent and follow verbal and written instructions in English.

Exclusion Criteria:

* Type 1 or type 2 diabetes mellitus diagnosed according to American Diabetes Association criteria
* Unstable heart disease as evidenced by ongoing angina
* Congestive heart failure
* Uncontrolled hypertension (BP greater than 170/100 mmHg on or off antihypertensive medication)
* Uncontrolled dyslipidemia (LDL greater than 200 or TG greater than 400 on or off lipid lowering medication)
* Tobacco, marijuana, cocaine, or intravenous drug use
* Shift workers (night shift or alternating day/night shifts)
* Gastroparesis
* Inflammatory bowel disease or irritable bowel syndrome
* Malignancy treated with chemotherapy within the past 3 years
* History of pancreatitis
* Depression requiring hospitalization or diagnosis of psychosis
* Renal insufficiency (eGFR less than 50)
* Transaminases greater than 2 times above the normal range
* Pregnancy within 6 months of the screening visit
* Lactation
* Failure to use medically approved contraceptive methods (monophasic oral contraception, intra uterine device, surgical sterilization or 2 combined barrier methods)
* History of an eating disorder (anorexia, bulimia or laxative abuse)
* Treatment with FDA-approved or over-the-counter weight loss medication within 6 months, with the exception of Xenical if there was no weight loss
* History of gastric bypass surgery or gastric stapling
* Biochemical evidence of hyper or hypothyroidism, or new diagnosis of hypo or hyperthyroidism within 3 months of screening visit
* Previous treatment with exenatide
* Discretion of the PI

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 249 (Actual)
Dates: Start 2012-03; Primary Completion 2019-01 (Actual); Study Completion 2019-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eleftheria Maratos-Flier, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rodgers M, Migdal AL, Rodriguez TG, Chen ZZ, Nath AK, Gerszten RE, Kasid N, Toschi E, Tripaldi J, Heineman B, Phan M, Ngo L, Maratos-Flier E, Dushay J. Weight Loss Outcomes Among Early High Responders to Exenatide Treatment: A Randomized, Placebo Controlled Study in Overweight and Obese Women. Front Endocrinol (Lausanne). 2021 Nov 17;12:742873. doi: 10.3389/fendo.2021.742873. eCollection 2021. PMID 34867786

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 249 subjects provided informed consent, 182 were randomized. I am reporting that 249 subjects were enrolled according to our local IRB definition of enrollment. 182 started study treatment. 67 subjects who did not start treatment were either found to be ineligible based on screening labs; withdrew consent; or were lost to followup.
Groups:
- Exenatide; Placebo: Subjects will be randomly assigned to the exenatide study treatment group or to the placebo study treatment group.
  Subjects will inject 5mcg of exenatide or identically dispensed placebo subcutaneously 15 minutes before the morning and evening meal for the first 2 weeks of the study. At study week 2, subjects will increase to 10mcg twice daily for the remainder of the study.
Period: Overall Study
Arm/Group | Exenatide | Placebo
Started | 127 | 55
Completed | 75 | 33
Not Completed | 52 | 22
Not completed — Lost to Follow-up | 20 | 8
Not completed — Withdrawal by Subject | 21 | 11
Not completed — Adverse Event | 11 | 3

BASELINE CHARACTERISTICS:
Population: Analysis population is the same as baseline population
Groups:
- Exenatide: Subjects will be randomly assigned to the exenatide study treatment group or to the placebo study treatment group.
  Exenatide: Subjects will inject 5mcg of exenatide or identically dispensed placebo subcutaneously 15 minutes before the morning and evening meal for the first 2 weeks of the study. At study week 2, subjects will increase to 10mcg twice daily for the remainder of the study.
- Placebo: Subjects will be randomly assigned to the exenatide study treatment group or to the placebo study treatment group.
  Placebo: Subjects will inject 5mcg of exenatide or identically dispensed placebo subcutaneously 15 minutes before the morning and evening meal for the first 2 weeks of the study. At study week 2, subjects will increase to 10mcg twice daily for the remainder of the study.
  Dietary counseling: All subjects will also receive individualized dietary counseling. Subjects may or may not be asked to follow a reduced calorie diet in addition to receiving treatment.
- Total: Total of all reporting groups
Arm/Group | Exenatide | Placebo | Total
Number analyzed (Participants) | 127 | 55 | 182
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.9 (11.9) | 44.6 (13.7) | 44.2 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 127 | 55 | 182
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 18 | 4 | 22
  Not Hispanic or Latino | 109 | 51 | 160
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 33 | 11 | 44
  White | 92 | 41 | 133
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 127 | 55 | 182

OUTCOME MEASURES:

1. Primary Outcome: Change in Body Weight
Description: Change in body weight after 12 weeks of treatment with exenatide or placebo twice daily injections. This outcome compares baseline and 12 week body weight.
Time Frame: 12 weeks
Population: subjects randomized to exenatide or placebo
Measure: Mean (Standard Deviation); unit: percentage weight loss
Arm/Group | Exenatide | Placebo
Number analyzed (Participants) | 75 | 33
percentage weight loss | 6.5 (0.4) | 7.5 (0.6)
Statistical Analysis 1: Comparison: Exenatide vs Placebo; Test type: Superiority; p < 0.05, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Entire study duration, up to 1 year
Description: Adverse events and serious adverse events are defined according to clinicaltrials.gov definition. Adverse event information was collected at each study visit, in person.
Groups:
- Exenatide: Exenatide: Subjects will inject 5mcg of exenatide or identically dispensed placebo subcutaneously 15 minutes before the morning and evening meal for the first 2 weeks of the study. At study week 2, subjects will increase to 10mcg twice daily for the remainder of the study.
- Placebo: Placebo: Subjects will inject 5mcg of exenatide or identically dispensed placebo subcutaneously 15 minutes before the morning and evening meal for the first 2 weeks of the study. At study week 2, subjects will increase to 10mcg twice daily for the remainder of the study.
  Dietary counseling: All subjects will also receive individualized dietary counseling. Subjects may or may not be asked to follow a reduced calorie diet in addition to receiving treatment.
Arm/Group | Exenatide | Placebo
All-Cause Mortality (participants affected / at risk) | 0/127 | 0/55
Serious Adverse Events (participants affected / at risk) | 0/127 | 0/55
Other Adverse Events (participants affected / at risk) | 89/127 | 14/55
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Exenatide (N=127) | Placebo (N=55)
nausea (Gastrointestinal disorders) | 89 | 14
diarrhea (Gastrointestinal disorders) | 24 | 9
vomiting (Gastrointestinal disorders) | 16 | 1
reflux (Gastrointestinal disorders) | 20 | 9
headache (Nervous system disorders) | 34 | 13
decreased appetite (Metabolism and nutrition disorders) | 52 | 13
rash (Skin and subcutaneous tissue disorders) | 14 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2018-01-09): https://cdn.clinicaltrials.gov/large-docs/33/NCT01590433/Prot_SAP_ICF_000.pdf